CLINICAL TRIAL: NCT07245017
Title: Randomized, Double-Blind, Placebo-Controlled, Single Center Clinical Trial to Evaluate the Safety and Preliminary Efficacy of JN002 Ophthalmic Solution in Adult Patients With Dry Eye Disease
Brief Title: JN002 for the Treatment of Dry Eye Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EENTFudan-JN002
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Placebo ophthalmic solution
  Interventions: Drug: Placebo Ophthalmic Solution (Vehicle)
- Low-Dose JN002 Group (Experimental): JN002 Ophthalmic Solution at a concentration of 0.05 mg/mL
  Interventions: Drug: JN002 Ophthalmic Solution (0.05 mg/mL)
- High-Dose JN002 Group (Experimental): JN002 Ophthalmic Solution at a concentration of 0.1 mg/mL
  Interventions: Drug: JN002 Ophthalmic Solution (0.1 mg/mL)

INTERVENTIONS:
Drug: Placebo Ophthalmic Solution (Vehicle) — Placebo ophthalmic solution (vehicle without active ingredient JN002), administered three times daily (1 drop per eye per dose) for 28 ± 2 consecutive days
  Arms: Placebo Group
Drug: JN002 Ophthalmic Solution (0.05 mg/mL) — JN002 Ophthalmic Solution at a concentration of 0.05 mg/mL, administered three times daily (1 drop per eye per dose) for 28 ± 2 consecutive days
  Arms: Low-Dose JN002 Group
Drug: JN002 Ophthalmic Solution (0.1 mg/mL) — JN002 Ophthalmic Solution at a concentration of 0.1 mg/mL, administered three times daily (1 drop per eye per dose) for 28 ± 2 consecutive days
  Arms: High-Dose JN002 Group

SUMMARY:
This is a first-in-human, single-center, randomized, double-blind, placebo-controlled clinical trial designed to:·Evaluate the efficacy of JN002 Ophthalmic Solution in treating dry eye disease (DED)·Assess the safety of JN002 Ophthalmic SolutionResearchers will compare three groups-placebo (vehicle), low-dose JN002 (0.05 mg/mL), and high-dose JN002 (0.1 mg/mL)-to evaluate whether JN002 Ophthalmic Solution improves DED outcomes and to assess its safety profile relative to placebo.Participants will:·Complete a baseline assessment (V0) including ocular exams, OSDI questionnaire, and systemic evaluation;·Administer the assigned study medication three times daily (1 drop per eye per administration);·Attend three follow-up visits (V1: 7±2 days, V2: 14±2 days, V3: 28±2 days post-treatment initiation) for ocular assessments, symptom queries, and adherence checks;·Undergo a full repeat of baseline assessments at V3 to evaluate treatment effects and safety profile

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Ocular Surface Disease Index (OSDI) score ≥ 13
3. Schirmer I test result ≤ 10 mm/5 min
4. Fluorescein tear film break-up time < 10 seconds
5. Corneal Fluorescein Staining score (National Eye Institute grading) ≥ 4
6. Best corrected visual acuity ≥ 0.6
7. Intraocular pressure ≤ 21 mmHg
8. Voluntarily agrees to participate in the study

Exclusion Criteria:

1. History of refractive surgery or intraocular surgery within the past 6 months
2. Clinically relevant ocular abnormalities at screening or baseline, including but not restricted to eye trauma, pterygium, allergic keratoconjunctivitis, active ocular infections, or abnormal ocular structures
3. Uncontrolled ocular or systemic diseases
4. Other conditions deemed by the investigators likely to interfere with study parameters
5. Females with plans for pregnancy at enrollment or during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining score | Baseline, 7±2 days, 14±2 days and 28 ± 2 days
  Change from baseline in Corneal Fluorescein Staining (CFS) score at the 7±2 days, 14±2 days and 28±2 days follow-up. CFS is evaluated following the guidelines from the National Eye Institute: the corneal surface is divided into five regions (central, superior, inferior, nasal, temporal), with each region assigned a score ranging from 0 to 3, resulting in a total possible score of 0 to 15-higher scores indicate more severe corneal epithelial damage and a worse clinical outcome.
Ocular Surface Disease Index score | Baseline, 7±2 days, 14±2 days and 28±2 days
  Change from baseline in Ocular Surface Disease Index (OSDI) score at the 7±2 days, 14±2 days and 28±2 days follow-up. OSDI is assessed via a 12-item self-reported questionnaire, where raw scores are converted to a standardized 0-100 scale through a specific calculation, with higher scores indicating more severe ocular surface disease symptoms.

SECONDARY OUTCOMES:
Schirmer I test | Baseline and 28 ± 2 days
  Change from baseline in Schirmer I test result (measuring aqueous tear secretion) at the 28±2 days follow-up.
Tear meniscus height | Baseline and 28 ± 2 days
  Change from baseline in tear meniscus height at the 28±2 days follow-up.
Non-invasive tear film break-up time | Baseline and 28 ± 2 days
  Change from baseline in non-invasive tear film break-up time (measured via Keratograph 5M) at the 28±2 days follow-up.
Tear inflammatory cytokines | Baseline and 28 ± 2 days
  Change from baseline in tear inflammatory cytokines (IL-1β, IL-6, IL-17A, TNF-α, INF-γ) levels at the 28±2 days follow-up.

OTHER OUTCOMES:
Corneal dendritic cell density | Baseline and 28 ± 2 days
  Change from baseline in corneal dendritic cell density at the 28±2 days follow-up, assessed and quantified via in vivo corneal confocal microscopy (IVCM)-a specialized imaging tool for ocular surface evaluation.
Best-corrected visual acuity | Baseline, 7 ± 2 days, 14 ± 2 days, and 28 ± 2 days
  Best-corrected visual acuity assessed at baseline, 7±2 days, 14±2 days, and 28±2 days.
Intraocular pressure | Baseline, 7±2 days, 14±2 days, and 28±2 days.
  Intraocular pressure assessed at baseline, 7±2 days, 14±2 days, and 28±2 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No